CLINICAL TRIAL: NCT01191931
Title: Prostate HistoScanning for the Non-invasive Detection and Staging of Prostate Cancer and Characterization of Prostate Tissues (PHS-02)
Acronym: PHS-02
Status: Completed | Type: Observational
Sponsor: Advanced Medical Diagnostics s.a. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR2P00113
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — paraffin blocks of prostate specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- prostate cancer: Patients with histologically proven prostate cancer (positive biopsy) and who are planned to undergo radical prostatectomy.

SUMMARY:
Study design:

-The study will be a phase I like study to assess the extent to which prostate HistoScanning (PHS, the index test) can identify and characterize foci of prostate cancer when compared to histological samples harvested during radical prostatectomy (the reference test). The study will comprise 3 steps: first, defining the most suitable method for matching the TRUS (TransRectalUltrasonography) to histology (step 1); second, refining the algorithms (training set); third, verification of the PHS performances (test set).

Study objectives:

* Primary Objective:

  * To evaluate the extent to which PHS can discriminate between malignant lesions of the prostate versus non-malignant tissue in 3D RF TRUS data using radical prostatectomy histological step sectioning as the reference test.
* Secondary Objectives:

  * To adapt and refine PHS tissue characterisation algorithms using RF data that were previously developed using grey-level data as input.
  * To assess the accuracy of PHS in predicting the volume of prostate cancers determined by histology.
  * To assess the ability of PHS to rule in or rule out the presence of cancer > or = 0.5 cc and of > or = 0.2 cc as determined by histology.
  * To evaluate the ability to discriminate primary Gleason pattern 4 and 5 versus 3 or less in tumours > or = 0.5 cc and > or = 0.2 cc.
  * To assess the ability of PHS to correctly risk stratify patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: >or=18 year-old
* Histologically (positive biopsy) proven prostate cancer with primary and secondary Gleason patterns attributed.
* Patient planned to undergo radical prostatectomy
* Prostate cancer is deemed to be organ confined (T1-T2, Nx or No, Mx or Mo)
* No prior treatment for prostate cancer, including any type of hormonal therapy
* No major calcification is noted during the TRUS (i.e. (Diameter >or=5 mm, spread all over the prostate or blocking to much of the ultrasound signal).
* Patient willing to give written informed consent

Exclusion Criteria:

* Patients who are either unsuitable or unwilling to enter the study or to proceed to surgical investigation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven prostate cancer (positive biopsy) and who are planned to undergo radical prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-02; Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Bleiberg, MD, Study Director
Locations (7):
- Belgium (2):
  - Bordet Institute, Brussels, Brussels Capital
  - UZ-Brussel, Brussels, Brussels Capital
- Olomouc Hospital, Olomouc, Czechia
- Universitätsklinikum Tübingen, Tübingen, Tübingen, Germany
- Semmelweis University, Budapest, Budapest, Hungary
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, Hammersmith, London
  - University College London Hospital (UCLH), London

REFERENCES:
- [Background] Braeckman J, Autier P, Garbar C, Marichal MP, Soviany C, Nir R, Nir D, Michielsen D, Bleiberg H, Egevad L, Emberton M. Computer-aided ultrasonography (HistoScanning): a novel technology for locating and characterizing prostate cancer. BJU Int. 2008 Feb;101(3):293-8. doi: 10.1111/j.1464-410X.2007.07232.x. Epub 2007 Oct 8. PMID 17922870
- [Background] Braeckman J, Autier P, Soviany C, Nir R, Nir D, Michielsen D, Treurnicht K, Jarmulowicz M, Bleiberg H, Govindaraju S, Emberton M. The accuracy of transrectal ultrasonography supplemented with computer-aided ultrasonography for detecting small prostate cancers. BJU Int. 2008 Dec;102(11):1560-5. doi: 10.1111/j.1464-410X.2008.07878.x. Epub 2008 Aug 14. PMID 18710457
- [Background] Lucidarme O, Akakpo JP, Granberg S, Sideri M, Levavi H, Schneider A, Autier P, Nir D, Bleiberg H; Ovarian HistoScanning Clinical Study Group. A new computer-aided diagnostic tool for non-invasive characterisation of malignant ovarian masses: results of a multicentre validation study. Eur Radiol. 2010 Aug;20(8):1822-30. doi: 10.1007/s00330-010-1750-6. Epub 2010 Mar 20. PMID 20306081
- [Background] Vaes E, Manchanda R, Nir R, Nir D, Bleiberg H, Autier P, Menon U, Robert A. Mathematical models to discriminate between benign and malignant adnexal masses: potential diagnostic improvement using ovarian HistoScanning. Int J Gynecol Cancer. 2011 Jan;21(1):35-43. doi: 10.1097/IGC.0b013e3182000528. PMID 21330829
- [Background] Salomon G, Spethmann J, Beckmann A, Autier P, Moore C, Durner L, Sandmann M, Haese A, Schlomm T, Michl U, Heinzer H, Graefen M, Steuber T. Accuracy of HistoScanning for the prediction of a negative surgical margin in patients undergoing radical prostatectomy. BJU Int. 2013 Jan;111(1):60-6. doi: 10.1111/j.1464-410X.2012.11396.x. Epub 2012 Aug 9. PMID 22882794
- [Result] Simmons LA, Autier P, Zat'ura F, Braeckman J, Peltier A, Romic I, Stenzl A, Treurnicht K, Walker T, Nir D, Moore CM, Emberton M. Detection, localisation and characterisation of prostate cancer by prostate HistoScanning(). BJU Int. 2012 Jul;110(1):28-35. doi: 10.1111/j.1464-410X.2011.10734.x. Epub 2011 Nov 17. PMID 22093966